CLINICAL TRIAL: NCT05852249
Title: Neutrocheck Summative Usability Study
Brief Title: Investigation of the Usability of Neutrocheck Amongst Healthy Volunteers and Healthcare Professionals.
Acronym: NeutroUSE
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: 52 North Health Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: NeutroUSE
Record Dates: First submitted 2023-04-19; First posted 2023-05-10 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-05

CONDITIONS: Neutropenia; Neutropenia, Febrile; Neutropenic Sepsis (Disorder)
MeSH Terms: conditions — Neutropenia; Febrile Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Paper instruction: Participants in this group will use paper instructions to use Neutrocheck.
- App instruction: Participants in this group will use App instructions to use Neutrocheck.

SUMMARY:
This study proposes to assess the usability of the Neutrocheck device and test kit amongst healthy volunteers and healthcare professionals (HCPs).

Neutrocheck is a portable, single-use diagnostic test intended to aid the diagnosis of neutropenia, febrile neutropenia and neutropenic sepsis using a finger prick blood sample.

Neutropenia is when the number of infection-fighting neutrophil cells in the blood are lower than normal. It can be caused by treatments such as chemotherapy or by certain medical conditions. Neutropenic sepsis is a life-threatening medical emergency that occurs when patients with neutropenia develop an infection. There is currently no way to test for neutropenic sepsis outside of hospitals. Neutrocheck is being developed for use as a self-test by patients at home alongside remote consultation with a HCP or at point-of-care by a HCP. This will allow rapid identification of patients requiring urgent intravenous antibiotics and medical assessment. In cases where Neutrocheck has eliminated the possibility of neutropenic sepsis, patients can avoid unnecessary and stressful hospital visits and valuable hospital resources will be saved.

Participants in this study will be invited to use the Neutrocheck test kit in a setting similar to a home environment to carry out a test, whilst being observed by a study moderator.

The Neutrocheck devices used in the study will be for investigational use only. This study will not be testing the accuracy of the Neutrocheck result, rather if Neutrocheck can be used safely and in a user-friendly way. Results will not be considered valid. Planned study duration is 2 months. This approach will enable us to complete the current phase of development and advance to a clinical validation study of Neutrocheck, assessing the diagnostic accuracy of Neutrocheck amongst users including those at risk of neutropenia and neutropenic sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent to participate
* Age 18 years or over

Exclusion Criteria:

* Known HIV or active Hep B or Hep C infection
* Phobia of needles or blood
* Currently undergoing immunosuppressive medical treatment or have received immunosuppressive treatment in the previous 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Identification of use errors, close calls and use difficulties associated with selected hazard-related use scenarios and participant's perceived root causes of these. | 2 months
Administration of a questionnaire to assess the effectiveness of key information for safety. | 2 months
  Participants will be asked to complete a questionnaire consisting of multiple choice questions related to key safety information for use of Neutrocheck. For example, this includes questions on storage of the device, expiry date and when to contact a healthcare professional. The data collected from the questionnaire will be summarised using descriptive statistics.

SECONDARY OUTCOMES:
Administration of a questionnaire to measure user satisfaction with the use of Neutorcheck | 2 months
  Participants will be asked to complete a questionnaire consisting of interval questions related to user satisfaction following use of Neutrocheck. The data collected from the questionnaire will be summarised using descriptive statistics.
Comparison of descriptive statistics for task completion rates, measured through observation, between two study groups, one using paper instructions and the other using app instructions. | 2 months
  Fisher's exact test will be used to determine the statistical significance of the differences in mean values between the two groups. To perform this analysis, we will utilise a statistical software such as R.
Comparison of user satisfaction, measured through a questionnaire, between two study groups: one group using paper instructions and the other using app instructions. | 2 months
  Fisher's exact test will be used to determine the statistical significance of the differences in mean values of responses between the two study groups completing the questionnaire. To perform this analysis, we will utilise a statistical software such as R.